CLINICAL TRIAL: NCT05623436
Title: The Effect of Ventrogluteal Injection Training Provided With Virtual Reality Technology on Knowledge, Skill, Motivation, and Anxiety Levels of Student: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality Technology in Ventrogluteal Injection Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, SEVGI DOGAN, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ATATURKU-SEVGİ
Record Dates: First submitted 2022-11-01; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Nursing Caries; Nursing Education
Keywords: intramuscular injection; nursing; simulation; virtual reality; ventrogluteal injection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Ventrogluteal injection training given by virtual reality technology is effective in increasing the knowledge and skill levels of students. It also has an impact on students' motivation and anxiety levels.
  Intervention: Behavioral: Education
  Interventions: Behavioral: Nursing students will be trained through virtual reality.
- Control (No Intervention): Ventrogluteal injection training given by virtual reality technology doesn't effective in increasing the knowledge and skill levels of students. It also hasn't an impact on students' motivation and anxiety levels.

INTERVENTIONS:
Behavioral: Nursing students will be trained through virtual reality. — Nursing students will be trained through virtual reality.
  Arms: Experimental

SUMMARY:
Intramuscular injections are one of the nursing functions frequently used in clinical practice. Sites used for the purpose of intramuscular injection; dorsogluteal, ventrogluteal, deltoid region, vastus lateralis muscle and rectus femoris muscle . Intramuscular injections can cause many complications. The most important complication is sciatic nerve injury, which may occur as a result of injection especially in the dorsogluteal region. In order to prevent complications that may develop as a result of intramuscular injection, it should be emphasized that the ventrogluteal region should be preferred in the selection of intramuscular injection site and students should be provided with the necessary knowledge and skills regarding injection from this region. In nursing education, many different methods are used with technological developments. One of them is simulation applications. There are various types of simulation applications. One of these simulation applications is virtual reality technology.

The goal of this interventional research is to evaluate the effect of ventrogluteal injection training developed by researchers and given to students through virtual reality glasses.

DETAILED DESCRIPTION:
The universe of the study consisted of first-year students enrolled in the "Basic Nursing and Clinical Skills" course in the nursing Turkish undergraduate program of Atatürk University Faculty of Nursing in the spring semester of the 2021-2022 academic year. The sample of the study consisted of students who had the research criteria and agreed to participate in the research. Prior to the study, a priori power analysis was performed to determine the sample size in this study. In the power analysis, it was determined that the sample size should be 128, 64 interventional and 64 control, at a significance level of 0.05, with a confidence interval of 95%, for power of 80%. Considering the data losses, it was decided to collect data from a total of 142 students by including 10% reserve sample in this number.

Inclusion criteria:

* Have not received previous application training for intramuscular injection
* Lack of experience in administering intramuscular injections
* Participation in the theoretical lecture presentation on intramuscular injection given by the instructor in the course "Basic Nursing and Clinical Skills"
* Absence of a health condition that prevents him from wearing virtual reality glasses and performing the study (Advanced vision problem, vertigo problem, etc.)
* Have not taken the Fundamentals of Nursing or Basic Nursing Care and Clinical Skills course before
* Understand the questions in forms and scales
* Willingness to participate in the study.

Exclusion criteria:

* The student does not participate in at least one of the research phases
* Receive of the student practical training for intramuscular injection from another instructor during the research process.

Variables of the research:

* Dependent Variable: After the application training with virtual reality simulation and intramuscular injection model, the knowledge evaluation scores, skill evaluation scores, motivation levels and anxiety levels of the students are dependent on the research.
* Independent Variable: Virtual reality simulation and application training with intramuscular injection model are independent variables of the research.
* Control Variable: The knowledge evaluation scores of the students before the application training are the control variable of the research.

Data collection tools:

"Introductory Questionnaire Form", "Intramuscular Injection Application to the Ventrogluteal Region Information Evaluation Form", "Motivation Scale for Teaching Material", "Status Anxiety Inventory" were used in data collection.

* Introductory Questionnaire Form: The form prepared by the researcher includes 9 questions including sociodemographic characteristics of the students such as age, gender and information about ventrogluteal region injection
* Intramuscular Injection Application Information Evaluation Form in the Ventrogluteal Region: This form has been prepared by the researcher in line with the literature by taking expert opinions. The Information Evaluation Form is a form consisting of 22 propositions in total that students can answer as "True", "False" and "I do not know". The form contains an equal number of "True" and "False" propositions. The form contains propositions that measure knowledge for ventrogluteal injection. The lowest score from the form is 0 and the highest score is 22. High scores obtained from the scale indicate that the level of information of the students is high.
* Intramuscular Injection to the Ventrogluteal Region Application Skill Evaluation Form: This form was prepared by the researcher based on the literature by taking expert opinions in order to evaluate the students' ability to apply intramuscular injection to the ventrogluteal region. The form includes intramuscular injection steps to the ventrogluteal region. The form contains 33 trading steps. The lowest score to be obtained from the form is 0 and the highest score is 100. High scores obtained from the scale indicate that the level of skill of the students is high.
* Motivation Scale for Instructional Material: The Cronbach alpha value of this scale, which consists of 33 items, has no inverse propositions and is of the five-point likert type, was found to be 0.97. The highest score that can be obtained from the scale is 165, while the lowest score is 33 points. A high overall score means that their level of motivation for the teaching material is high.
* Situational Anxiety Inventory: Situational Anxiety Inventory, consists of a total of twenty items. In the Situational Anxiety Inventory, the answers are grouped under 4 headings: "None", "A little", "Many", "Completely". Scores from the scale range from 20-80. The high score received is the high anxiety; If the score is low, it means that the anxiety is low. The analysis of scores in order of percentage is done in a similar way. A low percentage rank indicates that anxiety is low; A high percentage rank indicates that anxiety is high. The average score range determined in the application of the scale is between 36-41.

Pre-Application Phase:

Pre-application was made to 6 students randomly selected from the universe who agreed to participate in the study. Students who participated in the pre-practice were not included in the actual implementation phase of the research.

Data collection: The data were collected in the spring semester of the 2021-2022 academic year. The necessary explanations were made to the students who formed the sample of the research and their consent was obtained. Students whose consent was obtained were asked to fill out the "Introductory Questionnaire Form" and the "Intramuscular Injection Application Evaluation Form in the Ventrogluteal Region". All students who filled out these forms were shown the "Intramuscular Drug Administration Skill Video". According to the results of the students' knowledge evaluation scores, intervention and control groups were determined by randomization.

* Determination of Research Groups by Randomization: Students who met the criteria for inclusion in the study, who volunteered to participate in the research, who participated in the theoretical course presentation on intramuscular injection given by the instructor of the course in the "Basic Nursing and Clinical Skills" course were selected by randomization (n= 142) and included in the study. In the study, stratified sampling method was used for sample selection. In order to ensure that the students constituting the sample had similar characteristics, the knowledge levels of the students were determined by using the "Intramuscular Injection Application Information Evaluation Form in the Ventrogluteal Region" prepared by the researcher by taking expert opinions. According to the level of knowledge of the students; It was stratified into three groups as low , medium and high. First, students in the same group (Low, medium or high) with equal scores were randomly assigned to the intervention and control groups by lottery, respectively. After the students with equal scores were assigned to the groups, the remaining students were randomized first within the group and then between the groups. An equal number of intervention (n=71) and control groups (n=71) were created.

The students, who were divided into intervention and control groups, participated in the training of intramuscular injection administration from the ventrogluteal region.

* The intervention group received its practical training with virtual reality glasses. In the training content, the procedure steps for intramuscular injection from the ventrogluteal region were explained and first shown 1 time by the researcher. Then, each of the researchers was enabled to practice with virtual reality glasses and the necessary feedback was made. Students who completed their education were asked to fill out the "Contract for Compliance with Student Research Rules" and "Motivation Scale for Teaching Material". After the training, an analysis session was held with the students.
* The control group performed the application training in intramuscular injection model. Later, the students participated in the practical training in groups of 5 people. The students in the control group were given the necessary training by the researcher on the intramuscular injection model by demonstration method. In the training content, the procedure steps for intramuscular injection from the ventrogluteal region were explained and first shown 1 time by the researcher. Then, each of the researchers was made to apply on the model and the necessary feedback was given. Students who completed their education were asked to fill out the "Contract for Compliance with Student Research Rules" and "Motivation Scale for Teaching Material".

After all students' practical training in both the experimental and control groups was over, an exam (Objective Structured Clinical Exam/OSCE) was conducted to determine the students' anxiety, knowledge and skill status. "Intramuscular Injection Application Information Evaluation Form for Ventrogluteal Region" and "Status Anxiety Inventory" were applied to the students. The skill status of the students was evaluated by the researcher and recorded in the "Intramuscular Injection Application Skill Evaluation Form in the Ventrogluteal Region".

After 1 month the 1st OSCE exam, students were subjected to the 2nd OSCE exam again. In this exam, which constitutes the follow-up stage, the procedures in the 1st OSCE exam were applied and evaluated by the researcher and recorded in the "Intramuscular Injection Application Skill Evaluation Form to the Ventrogluteal Region". In this exam, which constitutes the follow-up stage, the procedures in the 1st OSCE exam were applied and evaluated by the researcher and recorded in the "Intramuscular Injection Application Skill Evaluation Form to the Ventrogluteal Region".

Evaluation of the data:

In the evaluation of the data obtained from the research, the Statistical Package for Social Sciences (SPSS) 22.0 package program will be used. The normal distribution of the data will be looked at by the Shapiro Wilk test. Mean, standard deviation, median, min, max, number and percentages will be used to evaluate the data. In the comparison of the mean between two independent groups, if the variable is normally distributed, the independent sample t test; If it does not fall apart normally, Mann Whitney will be examined with a U test. In statistical comparisons, if the variable is normally distributed in the comparison of the mean between the two dependent groups, the paired sample t test; If it does not fall apart normally, it will be examined by Wilcoxon test. Chi-square test will be used in the comparisons between the two categorical groups. Statistical significance level will be accepted as p<0.05.

Difficulties and limitations of the study:

The limitation of this research is that it is carried out only with 1nd year nursing students studying at a university's nursing faculty.

ELIGIBILITY:
Inclusion Criteria:

* Have not received previous application training for intramuscular injection.
* Lack of experience in administering intramuscular injections.
* Participation in the theoretical lecture presentation on intramuscular injection given by the instructor in the course "Basic Nursing and Clinical Skills".
* Absence of a health condition that prevents him from wearing virtual reality glasses and performing the study (Advanced vision problem, vertigo problem, etc.).
* Have not taken the Fundamentals of Nursing or Basic Nursing Care and Clinical Skills course before.
* Understand the questions in forms and scales.
* Willingness to participate in the study.

Exclusion Criteria:

* The student does not participate in at least one of the stages of the research.
* Receive practical training for intramuscular injection from another instructor during the research process.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Intramuscular Injection Application to the Ventrogluteal Region Information Evaluation Form | 2 months
  The Information Evaluation Form is a form consisting of 22 propositions in total that students can answer as "True", "False" and "I do not know". The form contains an equal number of "True" and "False" propositions. The form contains propositions that measure knowledge for ventrogluteal injection. The lowest score from the form is 0 and the highest score is 22. High scores obtained from the scale indicate that the level of information of the students is high.
Intramuscular Injection to the Ventrogluteal Region Application Skill Evaluation Form | 2 months
  The form includes intramuscular injection steps to the ventrogluteal region. The form contains 33 trading steps. The lowest score to be obtained from the form is 0 and the highest score is 100. High scores obtained from the scale indicate that the level of skill of the students is high.

SECONDARY OUTCOMES:
Motivation Scale for Teaching Material | 1 month
  The Cronbach alpha value of this scale, which consists of 33 items, has no inverse propositions and is of the five-point likert type, was found to be 0.97. The highest score that can be obtained from the scale is 165, while the lowest score is 33 points. A high overall score means that their level of motivation for the teaching material is high.
Situational Anxiety Inventory | 2 months
  Situational Anxiety Inventory, consists of a total of twenty items. Scores from the scale range from 20-80. The average score range determined in the application of the scale is between 36-41. High scores obtained from the scale indicate that the level of anxiety of the students is high.

CONTACTS AND LOCATIONS:
Overall Officials: SEVGİ DOGAN, Study Director — ATATURK UNİVERSİTY
Locations (1):
- Atatürk University Faculty of Nursing, Department of Nursing Fundamentals, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Öner N, Le Compte A. Status and constant anxiety inventory handbook. Boğaziçi University Press. 1983; Istanbul.
- [Result] Dinçer S, Doğanay A. Motivation scale for teaching material (ÖMMÖ) Turkish Adaptation Study. Elementary Education Online, 2016; 15(4).